CLINICAL TRIAL: NCT07317635
Title: Impact of Implementing a National Classification of Surgical Emergencies on Postoperative Morbidity and Mortality: a Prospective Multicenter Observational Study After Implementation.
Acronym: CLASSES
Status: Not yet recruiting | Type: Observational
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-14
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Surgical Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before integration of classification of surgical emergencies: Before integration of classification of surgical emergencies
- After integration of classification of surgical emergencies: After integration of a classification of surgical emergencies with a cognitive aid
  Interventions: Other: Implementation of classification of surgical emergencies

INTERVENTIONS:
Other: Implementation of classification of surgical emergencies — Observation of practices prior and after implementation of classification of surgical emergencies
  Groups: After integration of classification of surgical emergencies

SUMMARY:
The ACUTE committee of the French Society of Anesthesia and Intensive Care (SFAR), in consultation with surgical societies, has developed a national classification of surgical emergencies to define the ideal time to surgery for each indication.

The goal is to integrate this classification with a cognitive aid to improve patient triage and reduce waiting times for emergency surgery.

This classification will be presented at the 2026 SFAR Congress and as a practical decision-making tool.

A prospective, multicenter study will then evaluate its impact by measuring the rate of severe postoperative complications at 30 days using the Comprehensive Complication Index (CCI).

The study will include 2500 patients over two-week periods between February and June 2027.

Expected benefits include reduced patient morbidity and hospital stay, along with better emergency surgery planning and standardization across healthcare centers.

DETAILED DESCRIPTION:
The ACUTE committee of the French Society of Anesthesia and Intensive Care (SFAR) has developed a national classification of surgical emergencies in consultation with all surgical societies to specify the ideal time before surgery for each surgical indication. The aim is to integrate this classification with a cognitive aid to help patients consider these timeframes, based on the surgical indication, and various other factors in order to improve triage and thus reduce waiting times before emergency surgery. This classification will be presented at the 2026 SFAR Congress, as well as in the form of a cognitive aid.

Main objective To evaluate the rate of severe postoperative complications, measured using the Clavien-Dindo score and continuously expressed using the Comprehensive Complication Index (CCI), at 30 days post-surgery after implementation of the national classification of surgical emergencies.

Methods This is a prospective, observational, multicenter study. The data collection period will consist of two consecutive weeks chosen by the inclusion center within the interval between February 1, 2027, and June 30, 2027. 100 patients will be included during each period per center, for a total of 2500 patients.

Expected outcomes and benefits of the study results for patients, public health, and public policy decisions.

For patients, reducing waiting times for emergency surgery is likely to decrease morbidity and mortality, serious complications, and length of hospital stay, while increasing the number of days spent at home and limiting reoperations and rehospitalizations.

For public health, the study will:

* document the organizational impact of national standardization;
* reduce inter-center variability;
* limit nighttime surgery;
* improve emergency surgical planning.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) undergoing non-cardiac emergency surgery, defined as surgery with a preoperative anesthetic consultation performed less than 48 hours before the surgical procedure.

Patient managed in a University Hospital (Centre Hospitalo-Universitaire) or General Hospital (Centre Hospitalier Général).

Patients must receive initial management and diagnosis in the emergency department of the investigating center.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults under legal protection (guardianship, curatorship, or judicial safeguard)
  Patients who object to the reuse of their personal data for research purposes
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative morbidity and mortality | At Day 30after surgery
  Postoperative morbidity and mortality assessed using the Clavien-Dindo score and expressed on a continuous scale by the Comprehensive Complication Index (CCI) at 30 days (D30)Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France